CLINICAL TRIAL: NCT03135691
Title: Intraoperative Ventilation Management and Postoperative Pulmonary Complications in Patients at High Risk for Obstructive Sleep Apnea
Brief Title: Intraop Ventilation Management and Postop Pulmonary Complications in High Risk Patients for OSA
Status: Withdrawn | Type: Observational
Why Stopped: unable to retrieve data from EMR.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kimmy Bais, Assistant Professor of Clinical Anesthesiology, Ohio State University
Other Study IDs: 2016H0423
Record Dates: First submitted 2017-01-30; First posted 2017-05-01 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at High Risk for OSA: Patients at High Risk for Obstructive Sleep Apnea Undergoing Laparoscopic Bariatric Surgery; retrospective study, no intervention administered.

SUMMARY:
Lung protective ventilation (LPV) has been proposed to reduce the incidence of postoperative pulmonary complications (PPCs), and protect against ventilator induced lung injury (VILI).

DETAILED DESCRIPTION:
LPV was first introduced in the intensive care units but has been recently adopted in the operating rooms. Obstructive sleep apnea (OSA) is a widely prevalent condition in obese patients and requires special attention in the operating room. Screening for OSA risk in surgical patients is a common practice. The STOP-BANG questionnaire is a common screening tool for OSA (Snoring, Tiredness, Observed apnea, high blood Pressure, BMI, Age, Neck circumference, and male Gender). The American Society of Anesthesiologists practice guidelines for the perioperative management of patients with OSA do not recommend any specific ventilation strategy to prevent PPCs in this population. To the knowledge of the investigators, the association between intraoperative ventilation strategies and PPCs in laparoscopic bariatric surgery patients, who have a high STOP-BANG score, has not been adequately investigated. The investigators propose a retrospective chart review of patients, 18 years of age and older, who underwent laparoscopic bariatric surgery, in reverse Trendelenburg position, using pressure controlled ventilation (PCV/PCV-VG) at the Ohio State University Wexner Medical Center, between January 01, 2012 and November 22, 2016, to determine whether intraoperative driving pressure is a predictor of postoperative pulmonary complications. No procedures will be done for the sake of conducting this study except for a retrospective review of patient charts. Preoperative and intraoperative variables will be collected to determine their predictive value of postoperative complications. No risks to the patients' health or well being are anticipated due to the conduct of the proposed study. No immediate benefits to the patients from whom data was collected is anticipated either. Results obtained from this study may provide valuable information on the preferred ventilation strategies in the operating room for future patients who have a high risk of postoperative lung complications.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age ≥ 18 y/o
* Patients who underwent laparoscopic bariatric surgery
* Surgery under general anesthesia with endotracheal intubation and pressure controlled mode of ventilation (PCV or PCV-VG)

Exclusion Criteria:

* Pregnant females, prisoners
* Short procedures: time of mechanical ventilation < 60 minutes
* Patients who received volume controlled ventilation (VCV) mode
* Patients with past medical history of neuromuscular illnesses, pulmonary hypertension or CHF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include patients 18 years of age and older who underwent laparoscopic bariatric surgery, in reverse Trendelenburg position, using pressure controlled ventilation (PCV/PCV-VG) at the Ohio State University Wexner Medical Center, between January 01, 2014 and December 07, 2016.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Post-Operative Pulmonary Complications | After surgery until 30 days
  Incidence of any post-operative pulmonary complications up to 30 days after surgery in patients at high risk for OSA undergoing laparoscopic bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Lindsey, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No